CLINICAL TRIAL: NCT02212873
Title: School-based Intervention Program - My Body is Fit and Fabulous
Brief Title: My Body is Fit and Fabulous at School
Acronym: MyBFF@school
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Wan Nazaimoon WM, Dr, Ministry of Health, Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR1343916563
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Overweight; Obese
Keywords: school based intervention; overweight; obese; BMI z score; fat mass
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Equal number of age-matched overweight and obese students will be selected from a control school. There will be no intervention, and students will participate in their usual health and physical education classes plus any other curriculum activities provided by the school.
- MyBFF@school program (Experimental): Students will participate in all 3 components of MyFF@school for a total of 32 weeks; 1-hour of SSG thrice weekly plus 30 to 45 minutes of either nutrition or psychology classes once a week. All students including those in the control arm will be assessed at baseline, week-16 and at end of the study. They will undergo anthropometric measurements, body fat assessment, clinical examination and fitness test by modified Harvard step-test.
  Interventions: Other: MyBFF@school program

INTERVENTIONS:
Other: MyBFF@school program — Students will be required to participate in all 3 components of MyBFF@school (SSG, nutrition and psychology sessions) for 16 weeks under the supervision of trained researchers, then for another 16 weeks supervised by their respective teachers-in-charge of physical education and/or co-curriculum activity. Each SSG session will be for an hour, thrice weekly while the nutrition or psychology session will be for 30-45 minutes once a week.
  Arms: MyBFF@school program

SUMMARY:
In order to address and curb the high prevalence of childhood obesity in Malaysia, a school-based intervention program, MyBFF@school is developed for implementation in all schools in the country. The program is specific for overweight and obese students and it is hypothesized that by participating in this program, students will be able to control their body mass index.

DETAILED DESCRIPTION:
A nationwide Nutrition Survey of Malaysian Children carried out between 2008-2009 among 3542 children aged from 6 months to 12 years showed a prevalence of 9.8% overweight and 11.8% obesity while in a more recent 2011 Global School-based Student Heath Survey showed that the percentage of overweight and obese Malaysian school children age 13-15 years old was 25.4% and 10.9% respectively . If left unchecked, these children will grow up to be obese adults, developed various obesity-related complications such as cardiovascular diseases, diabetes etc. Realising the urgent needs to address the problems, the Ministry of Health Malaysia with the cooperation of the Ministry of Education, proposed to implement MyBFF@school in all schools in Malaysia. Students participating in MyBFF@school will take part in a structured physical activity in the form of small sided football game (SSG), and are to attend intensified and interactive nutrition and psychology classes aimed at improving their knowledge, self-esteem and self-empowerment.

ELIGIBILITY:
Inclusion Criteria:

Classified as overweight and obese based on BMI of 85th percentile and above, according to WHO growth chart.

No medical conditions that could endanger their health when participating in MyBFF@school.

Obtained parental and assent consents.

Exclusion Criteria:

With either physical or mental disability. With medical condition that prevents him/her to participate in moderate-to-vigorous intensity physical activity.

With comorbidities that may interfere with the study such as diagnosed type 2 diabetes mellitus, hypertension, nephritic syndrome, epilepsy, congenital heart disease and skeletal anomalies.

On steroids, on anti-epileptics and on methylphenidate.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 332 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 32 weeks of intervention
  The primary outcome is reduction in the BMI z-score of participating students.

SECONDARY OUTCOMES:
Percentage body fat | 32 weeks of intervention
  Body fat of all participating students will be measured at baseline, week-16 and week-32 following intervention using Inbody 720 body composition analyzer (GE Healthcare).

CONTACTS AND LOCATIONS:
Overall Officials: Wan Nazaimoon Wan Mohamud, PhD, Principal Investigator — Institute for Medical Research, Ministry of Health Malaysia
Locations (1):
- SKPP/ SMK Presint 9(1), 9(2), 11(1), 14(1), Putrajaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Wan Mohd Zin RM, Jalaludin MY, Md Zain F, Hong JYH, Ahmad Kamil NZI, Mokhtar AH, Wan Mohamud WN. Lifestyle intervention improves cardiometabolic profiles among children with metabolically healthy and metabolically unhealthy obesity. Diabetol Metab Syndr. 2024 Nov 11;16(1):268. doi: 10.1186/s13098-024-01493-8. PMID 39523406